CLINICAL TRIAL: NCT01477996
Title: Pain After Intravitreal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Principal Investigator, Dr. Christiane I. Falkner-Radler, Principial investigator, The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FR-7-CI-2011
Record Dates: First submitted 2011-08-08; First posted 2011-11-23 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2011-11

CONDITIONS: Pain
Keywords: intravitreal therapy; pain scales; gauge; Pain Scores; Visual Analog Scale
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): 27-gauge needle
  Interventions: Procedure: 27-gauge
- Group 2 (Active Comparator): 30-gauge needle
  Interventions: Procedure: 30-gauge

INTERVENTIONS:
Procedure: 27-gauge — 27-gauge needle for IVT
  Arms: Group 1
Procedure: 30-gauge — 30-gauge needle for IVT
  Arms: Group 2

SUMMARY:
This randomized clinical trial is comparing two different needles (27 gauge versus 30 gauge) for intravitreal therapy (IVT). Standardized questionnaires and pain scales should allow for standard recommendation regarding the optimal needle size for IVT.

DETAILED DESCRIPTION:
Purpose: To evaluate the influence of the type of the needle on pain scores after intravitreal therapy (IVT).

Design: Randomized clinical trial Methods: A total of 200 patients, treated with an IVT for exudative age-related macular degeneration (AMD) or a vascular retinal disease, will be included and randomly assigned to be treated with either a 27-gauge needle (group 1) or a 30-gauge needle (group 2). After IVt the patient has to fill out a standardized questionnaire including pain scores on the visual analog scale after the surgical procedure.

Regression analysis of the scaled questionnaires should allow for a standard recommendation regarding the optimal needle size for minimal subjective pain during IVT.

ELIGIBILITY:
Inclusion Criteria:

* vitrearetinal disease including age-related macular degeneration,
* clinical significant macular edema due to diabetic retinopathy or other vascular disorders
* treatment with intravitreal therapy

Exclusion Criteria:

* missing informed consent
* age under 50 years

Min Age: 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Visual Analoge Scale | 1 day, after the intravitreal therapy (IVT)
  pain scores on the visual analog scale after the IVT

SECONDARY OUTCOMES:
patients demographic data | 1 day, record of patients data before or after intravitreal therapy (IVT)
  age, gender, number of IVT, surgeon, prior surgical procedures
Baker scale | 1 day, after the intravitreal therapy (IVT)
  pain scores on the baker scale after the IVT

CONTACTS AND LOCATIONS:
Overall Officials: Christiane I Falkner-Radler, MD, Principal Investigator — The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery; Susanne Binder, MD, Study Chair — The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Locations (1):
- The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery, Department of Ophthalmology; Rudolf Foundation Clinic, Juchgasse 25, Vienna, Austria